CLINICAL TRIAL: NCT03289130
Title: The North Carolina-Louisiana Prostate Cancer Project, Project 3 Ancillary Study
Brief Title: Dietary Factors and Racial Disparities in Prostate Cancer Aggressiveness
Acronym: PCaP
Status: Completed | Type: Observational
Sponsor: University of South Carolina (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of North Carolina, Chapel Hill (Other); Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Susan Steck, Associate Professor, University of South Carolina
Other Study IDs: DAMD-11-1-0568
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, serum, urine, adipose tissue, DNA extracted from whole blood, frozen tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The North Carolina-Louisiana Prostate Cancer Project is a population-based case-only study of over 2,000 men newly diagnosed with prostate cancer designed to address racial differences in prostate cancer aggressiveness and survival through a comprehensive evaluation of social, individual, and tumor level influences on prostate cancer aggressiveness. Project 3 specifically aims to examine nutritional modulation of prostate cancer aggressiveness using dietary assessment and biomarker-based data on dietary factors.

DETAILED DESCRIPTION:
A total of 2,258 (1,130 African Americans and 1128 European Americans) men newly diagnosed with prostate cancer in North Carolina and Louisiana were enrolled into the study between 2004 and 2009. Participants signed informed consent and were interviewed by a trained nurse who collected information on demographics, occupation, family history, health status, health care, prostate cancer diagnosis and screening history, medication use, anthropometrics, lifestyle factors (e.g., physical activity, smoking), and diet and supplement use. Research subjects were asked to recall their diet in the year prior to prostate cancer diagnosis via a modified version of the National Cancer Institute Diet History Questionnaire. Vitamin and supplement use in the year prior to prostate cancer diagnosis was assessed via a validated questionnaire, and current use was assessed by bottle label inventory. Blood, urine, and adipose tissue samples were collected.

ELIGIBILITY:
Inclusion Criteria:

* first diagnosis of histologically confirmed adenocarcinoma of the prostate
* 40-79 years old at diagnosis,
* can complete the study interview in English,
* do not live in an institution (nursing home),
* are not cognitively impaired or in a severely debilitated physical state,
* are not under the influence of alcohol, severely medicated, or apparently psychotic at the time of the interview.
* must self-identify as at least part African American/Black or Caucasian American/White/European American.

Exclusion Criteria:

-

Ages: 40 Years to 79 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Only males were enrolled (prostate cancer only occurs in males).
Study Population: Residents of North Carolina and Louisiana with a first diagnosis of prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2258 (Actual)
Dates: Start 2004-09 (Actual); Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
High aggressive prostate cancer | Baseline (cross-sectional study)
  Gleason score>=8, or PSA>20ng/ml, or Gleason score>7 and clinical stage T3-T4

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Steck, Principal Investigator — University of South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data may be requested from PCaP through a centralized data request process.
Supporting Information: Study Protocol
Time Frame: Data are currently available indefinitely.
URL: https://pcap.bioinf.unc.edu/

REFERENCES:
- [Background] Schroeder JC, Bensen JT, Su LJ, Mishel M, Ivanova A, Smith GJ, Godley PA, Fontham ET, Mohler JL. The North Carolina-Louisiana Prostate Cancer Project (PCaP): methods and design of a multidisciplinary population-based cohort study of racial differences in prostate cancer outcomes. Prostate. 2006 Aug 1;66(11):1162-76. doi: 10.1002/pros.20449. PMID 16676364
- [Derived] Steck SE, Omofuma OO, Su LJ, Maise AA, Woloszynska-Read A, Johnson CS, Zhang H, Bensen JT, Fontham ETH, Mohler JL, Arab L. Calcium, magnesium, and whole-milk intakes and high-aggressive prostate cancer in the North Carolina-Louisiana Prostate Cancer Project (PCaP). Am J Clin Nutr. 2018 May 1;107(5):799-807. doi: 10.1093/ajcn/nqy037. PMID 29722851
- Available data/document: Individual Participant Data Set — https://pcap.bioinf.unc.edu/